CLINICAL TRIAL: NCT03641989
Title: Correlation Between Oral Health and Systemic Inflammation (COHESION)
Acronym: COHESION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshfield Clinic Research Foundation (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Amit Acharya, BDS, MS, PhD, Executive Director, Marshfield Clinic Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACH10317
Record Dates: First submitted 2018-06-26; First posted 2018-08-22 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Inflammation; Periodontal Disease; Gingivitis
Keywords: Toothpaste; Inflammation; Periodontal Disease; hsCRP; Oral health; Oral hygiene
MeSH Terms: conditions — Inflammation; Periodontal Diseases; Gingivitis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to brush twice daily for 30 days with the plaque disclosing agent toothpaste or a reference, non-plaque disclosing toothpaste. Toothpastes are comparable based on equivalent content of the active ingredient: fluoride.
Who Masked: Participant
Masking Description: Participants will not be told which toothpaste they have been given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plaque disclosing toothpaste (Active Comparator): Based on a randomization schema, a 30 day supply of the plaque disclosing toothpaste will be distributed to the participant. Participants will be instructed to brush two times a day for 30 days with the plaque disclosing toothpaste; avoiding the use of mouth rinses and floss. They will also be instructed to avoid any dental prophylaxis (e.g., cleaning, scaling or root planing to mechanically remove plaque and calculus) while on the trial and 30 days before they are enrolled.
  Interventions: Other: Plaque disclosing toothpaste
- Non-plaque disclosing toothpaste (Placebo Comparator): Based on a randomization schema, a 30 day supply of the over-the-counter, non-plaque disclosing toothpaste will be distributed to the participant. Participants will be instructed to brush two times a day for 30 days with the plaque disclosing toothpaste; avoiding the use of mouth rinses and floss. They will also be instructed to avoid any dental prophylaxis (e.g., cleaning, scaling or root planing to mechanically remove plaque and calculus) while on the trial and 30 days before they are enrolled.
  Interventions: Other: Non-plaque disclosing toothpaste

INTERVENTIONS:
Other: Plaque disclosing toothpaste — Plaque identifying toothpaste with a FDA-registered seed-extract dye (Annatto (Bixa Orellana)) and FD&C Blue No. 1.
  Arms: Plaque disclosing toothpaste
Other: Non-plaque disclosing toothpaste — Toothpaste that does not contain the FDA-registered seed-extract dye (Annatto (Bixa Orellana)) and FD&C Blue No. 1.
  Arms: Non-plaque disclosing toothpaste

SUMMARY:
COHESION is a randomized trial targeting reduction of systemic inflammation through an oral hygiene regimen incorporating a plaque-disclosing toothpaste and a control toothpaste.

DETAILED DESCRIPTION:
The present pilot trial will test the hypothesis that regular brushing with Plaque HD (interventional toothpaste) compared to conventional toothpaste (control) for 30 days in participants with confirmed mild to severe PD will significantly reduce hsCRP levels, a sensitive marker of inflammation and predictor of CVD. By completing the COHESION trial, we will collect important and relevant data to support application for investigator-initiated research funding from the US National Institutes of Health to directly test whether Plaque HD reduces CVD in larger, scaled multi-center randomized trial.

Participants will be asked to participate in three visits. During Visit One, we will be reviewing their medical and dental information as well as performing an oral evaluation to determine their level of gingivitis or periodontal disease. If the participant remains eligible, their blood will be drawn to determine whether the baseline hsCRP level falls within the eligible range (≥0.5 to ≤10.0 mg/L).

During Visit Two, if the participant remains eligible, they will be randomized and given a 30-day supply of the interventional or control toothpaste along with a study diary to track their progress.

The participant will receive a follow-up call 15 days after Visit Two to track compliance with study activity and monitor for any adverse events.

30-days later, during Visit Three, the participants will undergo another oral evaluation in addition to a second blood draw to measure the hsCRP level after using their assigned toothpaste for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Speak and understand English
* Willing and able to comply with all procedures for the duration of the trial
* ≥ 12 natural teeth
* Baseline hs-CRP level ≥0.5 and ≤10.0 mg/L
* No exposure to statins
* Presence of dental provider assessed gingivitis or mild, moderate or severe periodontitis based on the American Academy of Periodontology (AAP) and presence of visible plaque/calculus

Exclusion Criteria:

* Diagnosis or history of atherosclerosis, myocardial infarction, stroke, transient ischemic attack, peripheral vascular disease
* History of inflammatory conditions such as rheumatoid arthritis, lupus or other chronic inflammatory condition; cancer
* Exposure to statins
* Consistent or prescribed use of aspirin, nonsteroidal anti-inflammatory drugs (NSAIDS) or immunosuppressive drugs (defined as 10 or more doses in past 30 days)
* Removable appliances only if gum inflammation is present where the appliance is seated
* Dental prophylaxis [e.g., cleaning, scaling or root planning to mechanically remove plaque and calculus] within 30 days of randomization
* Infection anywhere in the body 2 weeks prior to baseline visit (excluding presence of PD) or exposure to antibiotics or anti-viral agents during this time frame
* Trauma to oral cavity within two weeks of baseline visit
* Current tobacco use
* Women who are pregnant or breast-feeding
* Use of any investigational products within 30 days of randomization
* History of allergies to dyes
* Deemed not suitable for study participation based on the clinical judgment of the investigator

Ages: 21 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in hsCRP levels with the use of the assigned toothpaste. | 30 days
  The primary outcome measure is magnitude of change in level of high sensitivity CRP (hsCRP) pre-trial compared to post trial as a surrogate marker to monitor change in local and systemic inflammation. Study eligible subjects with hsCRP levels between 0.5 and 10.0 mg/L at baseline (Visit 1) will be randomized to brushing for 30 days with one of two toothpastes followed by reassessment at visit 3 at the end of the intervention. Since distribution of hsCRP is skewed toward higher values, to satisfy statistical model assumptions, significance of the observed differences in outcomes between groups from baseline to day 30 will be tested on log-transformed data by using ANCOVA with treatment and baseline measurement as main factors and treatment by baseline measurement interaction. All significance tests for hsCRP will be conducted using R version 3.3.1 and two-sided significance levels of 0.05.

SECONDARY OUTCOMES:
Bleeding on Probing (BOP | 30 days
  Decrease in number of teeth with BOP following tooth-brushing intervention from baseline visit is a represents a primary clinical indicator of reduction in local inflammation of periodontal tissue. BOP per tooth will be evaluated by a dental professional using a periodontal probe along the gum line of each tooth at 6 sites per tooth at the baseline pre-trial visit (Visit One) and at post trial Visit Three after the 30 day tooth brushing intervention. The outcome measure will be the difference in the number of teeth exhibiting BOP pre and post the 30 day trial. This variable has no units and is a dichotomous nominal variable (i.e yes/no) evaluated on a per-tooth basis across total number of evaluable teeth present in the participant's mouth. (Scoring: 1=BOP present; 0=BOP absent).
Periodontal Pocket Depth (PPD) | 30 days
  PPD per tooth at 6 sites per tooth as a measure of periodontal health at baseline pre and post use of the assigned toothpaste will be assessed to determine presence and extent of PD. A dental professional will perform a periodontal assessment, pre (Visit one) and post (Visit three) the 30 day tooth brushing intervention applying Periodontology (AAP) 1999 Classification Criteria with 2015 updates to classify extent of PD as a continuous variable. PPD measurement, measured in mm, will be carried out pre and post clinical trial participation using a periodontal probe.
Plaque Levels | 30 days
  Each evaluable tooth will be examined by a dental professional for presence of supra-gingival biofilm deposited by oral pathogens using a periodontal probe at the pre baseline visit (Visit One) and post (Visit Three) visit following the 30 day tooth brushing intervention. Number of teeth with a change in visible plaque deposits post-trial compared to pre-trial levels will be determined. This variable has no units and will be evaluated as a dichotomous nominal variable (i.e., yes/no) on a per-tooth basis across total number of evaluable teeth. (Scoring: 1=visible plaque present; 0= no visible plaque).
Overall oral health assessment and analytical plan | 30 days
  Analytical plan for secondary outcomes: Significance of any differences in oral health characteristics at baseline (pre) and post intervention will be tested by t-tests for continuous and chi-square tests for discrete variables. For parameter estimation, means and mean ratios will calculated for each treatment group at each time point along with standard deviations. The purpose of collection of overall oral health assessment is to inform on the relative health of the participants mouth at time zero to support conduct of a sub-analysis to determine whether the magnitude of change in hsCRP correlated with relative health of the mouth determined during the pre-trial oral health assessment.
Evaluate CD4/CD8 ratio for participants over the age of 45 | 30 days
  CD4/CD8 ratios will be measured in the subset of subjects who meet eligibility based on hsCRP measures but whose CD4/CD8 ratio is less than 1.2 following analysis of blood collected in visit 1. Subjects whose CD4/CD8 ratio fell below 1.2 in visit 1 will have reassessment of CD4/CD8 ratio done on blood collected in visit 3. The magnitude of change in CD4/CD8 pre and post-trial will be evaluated tested by t-test analysis for this continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Acharya, BDS, MS, PhD, Principal Investigator — Marshfield Clinic Research Institute
Locations (1):
- Marshfield Clinic-Marshfield Center, Marshfield, Wisconsin, United States

REFERENCES:
- [Background] Eke PI, Dye BA, Wei L, Slade GD, Thornton-Evans GO, Borgnakke WS, Taylor GW, Page RC, Beck JD, Genco RJ. Update on Prevalence of Periodontitis in Adults in the United States: NHANES 2009 to 2012. J Periodontol. 2015 May;86(5):611-22. doi: 10.1902/jop.2015.140520. Epub 2015 Feb 17. PMID 25688694
- [Background] Glurich I, Acharya A, Shukla SK, Nycz GR, Brilliant MH. The oral-systemic personalized medicine model at Marshfield Clinic. Oral Dis. 2013 Jan;19(1):1-17. doi: 10.1111/j.1601-0825.2012.01921.x. Epub 2012 Mar 28. PMID 22458294
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Inflammation, aspirin, and the risk of cardiovascular disease in apparently healthy men. N Engl J Med. 1997 Apr 3;336(14):973-9. doi: 10.1056/NEJM199704033361401. PMID 9077376
- [Background] Demmer RT, Trinquart L, Zuk A, Fu BC, Blomkvist J, Michalowicz BS, Ravaud P, Desvarieux M. The influence of anti-infective periodontal treatment on C-reactive protein: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2013 Oct 14;8(10):e77441. doi: 10.1371/journal.pone.0077441. eCollection 2013. PMID 24155956
- [Background] Anitha V, Nair S, Shivakumar V, Shanmugam M, Priya BM, Rajesh P. Estimation of high sensitivity C-reactive protein in patients with periodontal disease and without coronary artery disease. Indian J Dent Res. 2015 Sep-Oct;26(5):500-3. doi: 10.4103/0970-9290.172048. PMID 26672420
- [Background] Ajwani S, Mattila KJ, Narhi TO, Tilvis RS, Ainamo A. Oral health status, C-reactive protein and mortality--a 10 year follow-up study. Gerodontology. 2003 Jul;20(1):32-40. doi: 10.1111/j.1741-2358.2003.00032.x. PMID 12926749
- [Background] VanWormer JJ, Acharya A, Greenlee RT, Nieto FJ. Oral hygiene and cardiometabolic disease risk in the survey of the health of Wisconsin. Community Dent Oral Epidemiol. 2013 Aug;41(4):374-84. doi: 10.1111/cdoe.12015. Epub 2012 Oct 29. PMID 23106415
- [Background] Fasula K, Evans CA, Boyd L, Giblin L, Belavsky BZ, Hetzel S, McBride P, DeMets DL, Hennekens CH. Randomized Trial of Plaque-Identifying Toothpaste: Decreasing Plaque and Inflammation. Am J Med. 2017 Jun;130(6):746-749. doi: 10.1016/j.amjmed.2016.09.003. Epub 2016 Oct 19. PMID 27771276
- [Background] Henson BS, Wong DT. Collection, storage, and processing of saliva samples for downstream molecular applications. Methods Mol Biol. 2010;666:21-30. doi: 10.1007/978-1-60761-820-1_2. PMID 20717775
- [Background] Lim Y, Totsika M, Morrison M, Punyadeera C. The saliva microbiome profiles are minimally affected by collection method or DNA extraction protocols. Sci Rep. 2017 Aug 17;7(1):8523. doi: 10.1038/s41598-017-07885-3. PMID 28819242
- See also: Wisconsin Department of Health Services. Deaths. — http://www.dhs.wisconsin.gov/stats/deaths/index.htm
- See also: Cornell University. Cardiovascular Disease in the United States: Economic Impacts — https://sites.google.com/a/cornell.edu/cardiovascular-disease-in-the-united-states/economic-impacts
- See also: Department of Health and Human Services (US). Sacher D. Oral health in America: a report of the Surgeon General. Rockville (MD): HHS, Office of the Surgeon General (US); 2000 — https://www.cdcfoundation.org/pr/2015/heart-disease-and-stroke-cost-america-nearly-1-billion-day-medical-costs-lost-productivity
- See also: Salimetrics. Saliva Collection and Handling Advice. 3rd Edition. 2015. — https://www.salimetrics.com/saliva-collection-handbook/